CLINICAL TRIAL: NCT00596817
Title: A Double-blind, Randomised, Placebo-controlled, Multicentre, Relapse-prevention Study With Two Doses of [Vortioxetine] Lu AA21004 in Patients With Major Depressive Disorder
Brief Title: Efficacy of Vortioxetine (Lu AA21004) in the Prevention of Relapse of Major Depressive Episodes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11985A; 2007-001871-13 (EudraCT Number)
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-02

CONDITIONS: Major Depressive Disorder
Keywords: Relapse prevention; Antidepressants; Placebo-controlled; Double-blind; Multicentre study
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Vortioxetine: 5 or 10 mg (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)

INTERVENTIONS:
Drug: Placebo — capsules, daily, orally
  Arms: Placebo
Drug: Vortioxetine (Lu AA21004) — encapsulated tablets, daily, orally
  Other Names: Brintellix
  Arms: Vortioxetine: 5 or 10 mg

SUMMARY:
This study will evaluate the efficacy of Vortioxetine in the prevention of relapse of major depressive episodes in patients who responded to open-label treatment with Vortioxetine.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Episode (MDE) as the primary diagnosis according to DSM-IV TR criteria
* At least one other MDE before the current one
* Moderate to severe depression

Exclusion Criteria:

* Any current psychiatric disorder other than Major Depressive Disorder (MDD) as defined in the DSM-IV TR
* Any substance disorder within the previous 6 months
* Female patients of childbearing potential who are not using effective contraception
* Use of any psychoactive medication 2 weeks prior to screening and during the study

Randomisation Criteria: Patients in remission (MADRS total score <=10) at both Week 10 and Week 12

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Result] Boulenger JP, Loft H, Florea I. A randomized clinical study of Lu AA21004 in the prevention of relapse in patients with major depressive disorder. J Psychopharmacol. 2012 Nov;26(11):1408-16. doi: 10.1177/0269881112441866. Epub 2012 Apr 9. PMID 22495621
- [Derived] Christensen MC, Florea I, Loft H, McIntyre RS. Efficacy of vortioxetine in patients with major depressive disorder reporting childhood or recent trauma. J Affect Disord. 2020 Feb 15;263:258-266. doi: 10.1016/j.jad.2019.11.074. Epub 2019 Nov 13. PMID 31818787
- [Derived] McIntyre RS, Florea I, Tonnoir B, Loft H, Lam RW, Christensen MC. Efficacy of Vortioxetine on Cognitive Functioning in Working Patients With Major Depressive Disorder. J Clin Psychiatry. 2017 Jan;78(1):115-121. doi: 10.4088/JCP.16m10744. PMID 27780334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were in- and outpatients from psychiatric settings.
Pre-assignment Details: The study consisted of two consecutive periods: a 12-week open-label treatment period with Vortioxetine and a double-blind, fixed-dose, placebo-controlled treatment period of at least 24 weeks.
Groups:
- Placebo: Placebo : capsules, daily, orally
- Vortioxetine: 5 or 10 mg: Vortioxetine (Lu AA21004) : encapsulated tablets, daily, orally
Period: Open-label Period
Arm/Group | Placebo | Vortioxetine: 5 or 10 mg
Started | 0 | 639
Completed | 0 | 492
Not Completed | 0 | 147
Not completed — Adverse Event | 0 | 49
Not completed — Lack of Efficacy | 0 | 33
Not completed — Other Reasons | 0 | 65
Period: Open-label Period to Double-blind Period
Arm/Group | Placebo | Vortioxetine: 5 or 10 mg
Started | 0 | 492
Completed | 0 | 400
Not Completed | 0 | 92
Not completed — Adverse Event | 0 | 5
Not completed — Lack of Efficacy | 0 | 24
Not completed — Not Eligible | 0 | 49
Not completed — Other Reasons | 0 | 14
Period: Double-blind Period
Arm/Group | Placebo | Vortioxetine: 5 or 10 mg
Started | 192 (194 patients were randomised. 2 did not receive study medication. 192 is full-analysis set (FAS).) | 204 (206 patients were randomised. 2 did not receive study medication. 204 is FAS.)
Completed | 104 | 125
Not Completed | 88 | 79
Not completed — Adverse Event | 5 | 16
Not completed — Lack of Efficacy | 52 | 28
Not completed — Non-compliance With Study Product | 3 | 4
Not completed — Protocol Violation | 11 | 8
Not completed — Withdrawal of Consent | 7 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Other Reasons | 10 | 18

BASELINE CHARACTERISTICS:
Population: The total number of patients under Baseline Measures is not 1035 as automatically calculated, but 639 as stated in the "Open-label Period (APTS)" column and 396 in the "Double-blind Period (FAS)".
  The "Total" column of each Baseline Measure is Double-blind Period (FAS).
Groups:
- Placebo - Double-blind Period (FAS): Placebo : capsules, daily, orally
- Vortioxetine: 5 or 10 mg - Double-blind Period (FAS): Vortioxetine (Lu AA21004) : encapsulated tablets, daily, orally
- Total: Total of all reporting groups
Arm/Group | Open-label Period (APTS) | Placebo - Double-blind Period (FAS) | Vortioxetine: 5 or 10 mg - Double-blind Period (FAS) | Total
Number analyzed (Participants) | 639 | 192 | 204 | 1035
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (12.4) | 45.1 (12.1) | 44.8 (12.4) | 45.0 (12.3)
Sex/Gender, Customized [Number; unit: participants]
  Female (Open-label Period) | 397 | NA — Only data for Open-label Period | NA — Only data for Open-label Period | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male (Open-label Period) | 242 | NA — Only data for Open-label Period | NA — Only data for Open-label Period | NA — Total not calculated because data are not available (NA) in one or more arms.
  Female (Double-blind Period) | 0 | 120 | 130 | 250
  Male (Double-blind Period) | 0 | 72 | 74 | 146
MADRS [Mean (Standard Deviation); unit: units on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
  units on a scale | 32.3 (4.1) | 4.66 (3.16) | 4.89 (3.00) | 4.78 (3.08)
HAM-D-17 [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Scale - 17 items (HAM-D-17) measures depression severity. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 52. The higher the score, the more severe.
  units on a scale | 22.8 (4.5) | 3.96 (3.15) | 4.46 (3.27) | 4.21 (3.21)
HAM-A [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56. The higher the score, the more severe.
  units on a scale | 22.6 (6.6) | 4.60 (3.60) | 5.09 (3.83) | 4.85 (3.72)
CGI-S [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
  units on a scale | 4.8 (0.7) | 1.54 (0.69) | 1.56 (0.68) | 1.55 (0.69)
SDS [Mean (Standard Deviation); unit: units on a scale] — The Sheehan Disability Scale (SDS) comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired). The higher the score, the more severe.
  units on a scale | 20.8 (5.7) | 8.37 (7.44) | 8.95 (7.09) | 8.66 (7.27)

OUTCOME MEASURES:

1. Primary Outcome: Relapse Within First 24 Weeks of the Double-blind Period Based on a MADRS Total Score >=22 or an Unsatisfactory Treatment Effect (Lack of Efficacy) as Judged by the Investigator
Description: The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
Time Frame: Within first 24 weeks of the double-blind period
Population: FAS
Measure: Number; unit: percentage of patients who relapsed
Groups:
- Vortioxetine: 5 or 10 mg: encapsulated tablets, daily, orally
Arm/Group | Placebo | Vortioxetine: 5 or 10 mg
Number analyzed (Participants) | 192 | 204
percentage of patients who relapsed | 26.0 | 13.2
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine: 5 or 10 mg; Test type: Superiority or Other; p = 0.0035, Cox-model; Cox-model using an exact method to handle ties; Hazard Ratio (HR) = 2.01, 95% CI 2-sided [1.26 to 3.21]

2. Secondary Outcome: Relapse During the Entire Double-blind Period Based on a MADRS Total Score >=22 or an Unsatisfactory Treatment Effect (Lack of Efficacy) as Judged by the Investigator
Time Frame: Within 64 weeks of the double-blind period
Population: FAS
Measure: Number; unit: percentage of patients who relapsed
Arm/Group | Placebo | Vortioxetine: 5 or 10 mg
Number analyzed (Participants) | 192 | 204
percentage of patients who relapsed | 30.2 | 15.2
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine: 5 or 10 mg; Test type: Superiority or Other; p = 0.0010, Cox-Model — A nominal p-value is provided; Hazard Ratio (HR) = 2.09, 95% CI 2-sided [1.35 to 3.23]

3. Secondary Outcome: Change From Double-blind Baseline in MADRS Total Score After 24 Weeks of Double-blind Treatment
Time Frame: Double-blind Baseline and Week 24 of the double-blind period
Population: FAS; observed cases (OC)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine: 5 or 10 mg
Number analyzed (Participants) | 132 | 151
units on a scale | 1.45 (0.55) | -0.62 (0.51)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine: 5 or 10 mg; Test type: Superiority or Other; p = 0.0020, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -2.06, 95% CI 2-sided [-3.36 to -0.77], Standard Error of Mean 0.66

4. Secondary Outcome: Change From Double-blind Baseline in HAM-D-17 Total Score After 24 Weeks of Double-blind Treatment
Description: The Hamilton Depression Scale - 17 items (HAM-D-17) measures depression severity. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 52. The higher the score, the more severe.
Time Frame: Double-blind Baseline and Week 24 of the double-blind period
Population: FAS; OC
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine: 5 or 10 mg
Number analyzed (Participants) | 136 | 158
units on a scale | 1.61 (0.46) | 0.30 (0.42)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine: 5 or 10 mg; Test type: Superiority or Other; p = 0.0171, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -1.31, 95% CI 2-sided [-2.39 to -0.24], Standard Error of Mean 0.55

5. Secondary Outcome: Change From Double-blind Baseline in HAM-A Total Score After 24 Weeks of Double-blind Treatment
Description: The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56. The higher the score, the more severe.
Time Frame: Double-blind Baseline and Week 24 of the double-blind period
Population: FAS; OC
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine: 5 or 10 mg
Number analyzed (Participants) | 136 | 158
units on a scale | 0.89 (0.50) | -0.23 (0.46)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine: 5 or 10 mg; Test type: Superiority or Other; p = 0.0612, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-2.30 to 0.05], Standard Error of Mean 0.60

6. Secondary Outcome: Change From Double-blind Baseline in CGI-S Score After 24 Weeks of Double-blind Treatment
Description: The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
Time Frame: Double-blind Baseline and Week 24 of the double-blind period
Population: FAS; OC
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine: 5 or 10 mg
Number analyzed (Participants) | 132 | 151
units on a scale | 0.24 (0.08) | -0.14 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine: 5 or 10 mg; Test type: Superiority or Other; p = 0.0002, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.57 to -0.18], Standard Error of Mean 0.10

7. Secondary Outcome: Proportion of Responders at Week 24 of the Double-blind Period (Response Defined as a >=50% Reduction in MADRS Total Score From Open-label Baseline)
Time Frame: Week 24 of the double-blind period (Counted From Open-label Baseline)
Population: FAS; OC
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Vortioxetine: 5 or 10 mg
Number analyzed (Participants) | 132 | 151
percentage of patients | 91.7 | 98.0
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine: 5 or 10 mg; Test type: Superiority or Other; p = 0.025, Fisher Exact — A nominal p-value is provided; Difference = 6.35, 95% CI 2-sided [1.13 to 11.56]

8. Secondary Outcome: Proportion of Remitters at Week 24 of the Double-blind Period (Remission Defined as a MADRS Total Score <=10)
Time Frame: Week 24 of the double-blind period
Population: FAS; OC
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Vortioxetine: 5 or 10 mg
Number analyzed (Participants) | 132 | 151
percentage of patients | 82.6 | 94.7
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine: 5 or 10 mg; Test type: Superiority or Other; p = 0.002, Fisher Exact — A nominal p-value is provided; Difference = 12.13, 95% CI 2-sided [4.73 to 19.52]

9. Secondary Outcome: Change From Double-blind Baseline in SDS Total Score at Week 24 of the Double-blind Period
Description: The Sheehan Disability Scale (SDS) comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired). The higher the score, the more severe.
Time Frame: Week 24 of the double-blind period (Counted From Double-blind Baseline)
Population: FAS; OC
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine: 5 or 10 mg
Number analyzed (Participants) | 118 | 135
units on a scale | 0.14 (0.58) | -0.53 (0.57)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine: 5 or 10 mg; Test type: Superiority or Other; p = 0.3642, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-2.12 to 0.78], Standard Error of Mean 0.73

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: 12-week open-label period, 24-week double-blind period and 4-week safety follow-up period. Other Adverse Events: 12-week open-label period and 24-week double-blind period.
Arm/Group | Open-label Period (APTS) | Placebo - Double-blind Period (FAS) | Vortioxetine: 5 or 10 mg - Double-blind Period (FAS)
Serious Adverse Events (participants affected / at risk) | 14/639 | 6/192 | 7/204
Other Adverse Events (participants affected / at risk) | 337/639 | 73/192 | 79/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Open-label Period (APTS) (N=639) | Placebo - Double-blind Period (FAS) (N=192) | Vortioxetine: 5 or 10 mg - Double-blind Period (FAS) (N=204)
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Sebaceous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Serotonin syndrome (Nervous system disorders) | 1 | 0 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0/397 | 0/120 | 1/130
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Social stay hospitalisation (Social circumstances) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Period (APTS) (N=639) | Placebo - Double-blind Period (FAS) (N=192) | Vortioxetine: 5 or 10 mg - Double-blind Period (FAS) (N=204)
Dry mouth (Gastrointestinal disorders) | 41 | 0 | 4
Nausea (Gastrointestinal disorders) | 164 | 6 | 18
Fatigue (General disorders) | 32 | 4 | 4
Gastroenteritis (Infections and infestations) | 12 | 6 | 11
Influenza (Infections and infestations) | 7 | 9 | 14
Nasopharyngitis (Infections and infestations) | 52 | 26 | 22
Accidental overdose (Injury, poisoning and procedural complications) | 36 | 15 | 16 — Everything beyond the prescribed dose, for instance one extra tablet, is counted as an overdose.
Dizziness (Nervous system disorders) | 44 | 7 | 6
Headache (Nervous system disorders) | 117 | 25 | 25
Insomnia (Psychiatric disorders) | 36 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The main publication has to be published before any sub-publications. H. Lundbeck A/S follows the Vancouver declaration with respect to authorship.